CLINICAL TRIAL: NCT00249236
Title: The Efficacy And Safety Of Flexible Dosage Ranges Of Risperidone Versus Placebo In The Treatment Of Manic Or Mixed Episodes Associated With Bipolar I Disorder
Brief Title: A Study of the Effectiveness and Safety of Risperidone Versus Placebo in the Treatment of Manic or Mixed Episodes Associated With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006064
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Bipolar Disorder; Manic Episode
Keywords: risperidone; antipsychotic agents; bipolar disorders; manic episode
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone, oral tablets

SUMMARY:
The purpose of the study is to assess the effectiveness and safety of risperidone (an antipsychotic medication) versus placebo in treating mania during 3 weeks of treatment in patients with Bipolar I Disorder who suffer from manic or mixed episodes.

DETAILED DESCRIPTION:
Antipsychotic agents have, for a long time, been used to alleviate the severe behavioral problems associated with manic episodes. Risperidone, widely used in the treatment of schizophrenia, has been shown to be effective in the treatment of manic and mixed episodes associated with bipolar disorders. This is a randomized, double-blind study to evaluate the effectiveness and safety of risperidone compared with placebo in the treatment of patients with bipolar disorder who are experiencing a manic or mixed episode. Patients who are voluntarily hospitalized at the time of study enrollment (for treatment of the manic episode) receive study medication to be taken orally, once a day. Patients receive placebo or risperidone at a starting dose of 3 mg, with gradual dose increases or decreases at the investigator's discretion within the daily dosing range of 1 to 6 mg to achieve optimal effectiveness, while minimizing any intolerance to the drug. Treatment with risperidone or placebo tablets continues for 3 weeks. The primary measure of efficacy is the change from baseline to the end of treatment in the Young Mania Rating Scale (YMRS); Other efficacy assessments include the changes in: the Clinical Global Impression-Severity of Illness (CGI-S) scale; Global Assessment Scale (GAS), which assesses the patient's level of functioning; and the Positive and Negative Syndromes Scale (PANSS), a scale for measuring psychotic symptoms. Safety assessments include the incidence of adverse events throughout the study; measurement of vital signs (temperature, pulse, blood pressure) and evaluation of the presence and severity of extrapyramidal symptoms by the Extrapyramidal Symptom Rating Scale (ESRS) at specified intervals; and clinical laboratory tests (hematology, biochemistry, urinalysis) at the start and end of the study. The study hypothesis is that daily treatment with risperidone is more effective than placebo, as measured by Young Mania Rating Scale scores, in the treatment of the manic phase of Bipolar I Disorder. Risperidone oral tablets, 1 mg, taken once daily in the evening; dose of 3 mg on Day 1; dose range of 2 - 4 mg on Day 2; dose range 1 - 5 mg on Day 3; dose range 1 - 6 mg on Days 4 - 21. Doses may be increased or decreased at investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for Bipolar I Disorder, Most Recent Episode Manic or Mixed
* hospitalized voluntarily at study initiation for treatment of manic episode
* history (prior to study initiation) of at least one documented manic or mixed episode that required treatment
* total score >=20 on the Young Mania Rating Scale (YMRS) at start of the study

Exclusion Criteria:

* Meets DSM-IV criteria for Schizoaffective Disorder or for rapid cycling
* borderline or antisocial personality disorder
* history of substance dependence (excluding nicotine and caffeine) within the 3 months prior to study initiation
* seizure disorder
* females who are pregnant or nursing, or those lacking adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2001-03; Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Change in Young Mania Rating Scale (YMRS) total score from baseline to end of treatment.

SECONDARY OUTCOMES:
Change from baseline to end of treatment in Clinical Global Impression-Severity of Illness (CGI-S) scale, Global Assessment Scale (GAS), and Positive and Negative Syndrome Scale (PANSS) total score; incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Khanna S, Vieta E, Lyons B, Grossman F, Eerdekens M, Kramer M. Risperidone in the treatment of acute mania: double-blind, placebo-controlled study. Br J Psychiatry. 2005 Sep;187:229-34. doi: 10.1192/bjp.187.3.229. PMID 16135859
- [Result] Gopal S, Steffens DC, Kramer ML, Olsen MK. Symptomatic remission in patients with bipolar mania: results from a double-blind, placebo-controlled trial of risperidone monotherapy. J Clin Psychiatry. 2005 Aug;66(8):1016-20. doi: 10.4088/jcp.v66n0809. PMID 16086617